CLINICAL TRIAL: NCT02258438
Title: Effect of Breaking up Prolonged Sitting on Metabolic Flexibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 14-0429; UL1TR001082 (NIH)
Record Dates: First submitted 2014-10-02; First posted 2014-10-07 (Estimated); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Health Behavior
Keywords: Sedentary Behavior
MeSH Terms: conditions — Health Behavior; Sedentary Behavior | interventions — Sitting Position

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Uninterrupted sitting (Experimental): Patient will refrain from any structured activity and reduce any daily life activity. The patient will spend 24 hours in the calorimeter room. During the 24 hours the patient will remain sedentary for the 24 hours but will be able to watch TV, computer work or read.
  Interventions: Behavioral: Uninterrupted sitting
- Sitting + 1 bout of activity (Experimental): The patient will be asked to perform the 45 minutes of moderate-exercise intervention in the morning once per day for two days in their daily life. This bout of exercise will be supervised by study staff on one of the treadmills On day 3 the patient will report at the Clinical and Translational Research Center (CTRC) of the University Hospital of Colorado and will spend 24hr in the room calorimeter. During the day, you will be asked to sit quietly in a chair, except to rise from the chair to void, and to perform one bout of 45-min moderate-intensity walking on a treadmill.
  Interventions: Behavioral: Sitting + 1 bout of activity
- Sitting + microbursts of activity (Experimental): The patient will be asked to refrain from any structured exercise running, swimming, lifting weights, yoga, dancing, etc.) for two days but to walk for the 5 minute intervention each hour between 1000 and 1800. On day 3, The patient will report at the CTRC of the University Hospital of Colorado and will spend 24hr in the room calorimeter. During the day, the patient will be asked to rise from the seated position every hour for 9 hours from 1000 to 1800 to complete 5 min moderate-intensity walking on a treadmill, which represents a total of 45 min.
  Interventions: Behavioral: Sitting + microbursts of activity

INTERVENTIONS:
Behavioral: Uninterrupted sitting — Subjects will be asked to refrain for two days from any structured activity and to reduce any daily life activity (walking, taking the stairs, biking, etc.) in their daily life. On day 3, subjects will remain seated all day in the room calorimeter, except to rise from the chair to void.
  Arms: Uninterrupted sitting
Behavioral: Sitting + 1 bout of activity — Subjects will be asked to perform 45 minutes of moderate-exercise in the morning once per day for two days in their daily life. On day 3 they will remain seated all day in the room calorimeter, except to rise from the chair to void, and to perform one bout of 45-min moderate-intensity (defined below) walking on a treadmill at 1000.
  Arms: Sitting + 1 bout of activity
Behavioral: Sitting + microbursts of activity — Subjects will be asked to refrain from any structured exercise for two days but to walk for 5 minutes each hour between 1000 and 1800 in daily life. On day 3, subjects will rise from the seated position every hour for 9 hours from 1000 to 1800 to complete 5min moderate-intensity (defined below) walking on a treadmill, which represents a total of 45min.
  Arms: Sitting + microbursts of activity

SUMMARY:
The investigators propose in this project to determine the effect of 3 days of frequent interruption of prolonged sitting on metabolic health in healthy overweight sedentary adults (n=24), as compared to 3 days including a single long bout of isocaloric exercise or a control condition where subjects do not exercise but are subjected to prolonged sitting. The investigators believe that this proposed project will provide an initial evidence base for the health benefits of breaking up prolonged sitting with short bursts of moderate-intensity activity, like walking.

DETAILED DESCRIPTION:
Although public-health recommendations to engage in moderate-to-vigorous physical activity (at least 30min, 5 days / week) have been widely promulgated by the government, most people are physically inactive. Sedentary behaviors, like time spent sitting, are associated with serious implications on metabolic health, indicating that even in individuals who regularly exercise a reduction in time spent sitting can confer health benefits. Encouraging recent evidence shows that walking breaks throughout the day are an effective strategy to offset the deleterious effects of prolonged uninterrupted sitting. Further data however are needed to better understand the effect of these microbursts of activity along the day. The investigators propose in this project to determine the effect of 3 days of frequent interruption of prolonged sitting on metabolic health in healthy overweight sedentary adults (n=24), as compared to 3 days including a single long bout of isocaloric exercise or a control condition where subjects do not exercise but are subjected to prolonged sitting. Plasma glucose, insulin, triglycerides and free fatty acids concentrations and the use of substrate (glucose, fat or protein) to provide energy to the body in response to meals consumption will be measured on day 3 of each of these three conditions. The investigators will furthermore assess the ability of the participants to perform the interventions on physical activity at the end of each day over the three days of intervention (2 days in free-living conditions and one day in a controlled environment). The investigators believe that this proposed project will provide an initial evidence base for the health benefits of breaking up prolonged sitting with short bursts of moderate-intensity activity, like walking. This innovative strategy may be more effective at combating the adverse effects of sedentary behaviors than more traditional approaches like structured exercise.

ELIGIBILITY:
Inclusion Criteria:

* overweight but weight stable (less than +/- 3kg over previous 6 months) male and female adults (n=24) will be recruited.
* age between 19-45 years old,
* a BMI of 27-33 kg/m2,
* inactive (≤ 1.5hr/wk of moderate-to-vigorous activity),
* sedentary (office employees who are spending more than 6hrs/day in sitting position) and
* English-speaking.

Exclusion Criteria:

* any history of renal, cardiovascular or hepatic diseases,
* type 1 or 2 diabetes,
* cancer,
* pregnancy,
* smoking,
* consumption of drugs or alcohol (>40g/d),
* any medications known to interfere with lipid or energy metabolism,
* known physical activity contraindications, or major illness/physical problems (acute or chronic) that may limit their ability to perform the walking activities and
* menopause (defined as no menses in the prior 6 months). The use of birth pill control will be accepted. Women are asked to avoid pregnancy until completion of Condition C.

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2014-10-08 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Total substrate oxidation | 1 day
  Total fat oxidation during the test day will be determined using whole-room indirect calorimetry. O2 consumption and CO2 production will be determined from the flow rates and differences in gas concentrations between air entering and air exiting the calorimeter as previously described
Postprandial plasma insulin and glucose response | 1 day
  Plasma glucose and insulin will be measured in fasting conditions and hourly during 12hrs following a standard meal consumption. The area under the curve will be calculated for both plasma glucose and insulin. This area will represent the postprandial response to a meal for both insulin and glucose.
Dietary fat oxidation | 1 day
  Subjects will collect their own hourly breath sampling for 13CO2 by blowing through a straw into two 15ml Vacutainer after the investigators will have shown them the procedure. Breath CO2 will be sampled directly from the Vacutainer with a syringe, and 13CO2 /12CO2 measured with Isotopic Ratio Mass Spectrometer (IRMS).

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Bergouignan, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Jong NP, Rynders CA, Goldstrohm DA, Pan Z, Lange AH, Mendez C, Melanson EL, Bessesen DH, Bergouignan A. Effect of frequent interruptions of sedentary time on nutrient metabolism in sedentary overweight male and female adults. J Appl Physiol (1985). 2019 Apr 1;126(4):984-992. doi: 10.1152/japplphysiol.00632.2018. Epub 2019 Jan 10. PMID 30629473